CLINICAL TRIAL: NCT05182840
Title: Randomised, Double-blind, Placebo-controlled and Parallel Dose Group Trial to Investigate Efficacy and Safety of Multiple Doses of Oral BI 690517 Over 14 Weeks, Alone and in Combination With Empagliflozin, in Patients With Diabetic and Non-diabetic Chronic Kidney Disease
Brief Title: A Study to Test Whether Different Doses of BI 690517 Alone or in Combination With Empagliflozin Improve Kidney Function in People With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1378.5; 2021-001434-19 (EudraCT Number); 1378-0005 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2022-01-05; First posted 2022-01-10 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Run-in period: 10 mg empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Run-in period: Placebo to empagliflozin 10 mg (Placebo Comparator)
  Interventions: Drug: Placebo to empagliflozin
- Treatment period: 10 mg empagliflozin + 3 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Empagliflozin
- Treatment period: 10 mg empagliflozin + 10 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Empagliflozin
- Treatment period: 10 mg empagliflozin + 20 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Empagliflozin
- Treatment period: 10 mg empagliflozin + Placebo to BI 690517 (Placebo Comparator)
  Interventions: Drug: Placebo to BI 690517; Drug: Empagliflozin
- Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo to empagliflozin
- Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo to empagliflozin
- Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 690517 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo to empagliflozin
- Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517 (Placebo Comparator)
  Interventions: Drug: Placebo to BI 690517; Drug: Placebo to empagliflozin

INTERVENTIONS:
Drug: BI 690517 — Film-coated tablets
  Other Names: Vicadrostat
  Arms: Treatment period: 10 mg empagliflozin + 10 mg BI 690517; Treatment period: 10 mg empagliflozin + 20 mg BI 690517; Treatment period: 10 mg empagliflozin + 3 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517
Drug: Placebo to BI 690517 — Film-coated tablets
  Arms: Treatment period: 10 mg empagliflozin + Placebo to BI 690517; Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517
Drug: Empagliflozin — Empagliflozin
  Arms: Run-in period: 10 mg empagliflozin; Treatment period: 10 mg empagliflozin + 10 mg BI 690517; Treatment period: 10 mg empagliflozin + 20 mg BI 690517; Treatment period: 10 mg empagliflozin + 3 mg BI 690517; Treatment period: 10 mg empagliflozin + Placebo to BI 690517
Drug: Placebo to empagliflozin — Placebo to empagliflozin
  Arms: Run-in period: Placebo to empagliflozin 10 mg; Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517; Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517

SUMMARY:
This study is open to adults with chronic kidney disease. People with and without type 2 diabetes can take part in this study.

The purpose of this study is to find out whether a medicine called BI 690517 improves kidney function in people with chronic kidney disease when taken alone or in combination with a medicine called empagliflozin.

In the first part of the study, participants take empagliflozin or placebo as tablets every day for 2 months. Placebo tablets look like empagliflozin tablets but do not contain any medicine.

In the second part, participants are divided into several groups. Depending on the group, the participants then additionally take different doses of BI 690517 or placebo as tablets for 3.5 months. In this case, placebo tablets look like BI 690517 tablets but do not contain any medicine.

Participants are in the study for about 6 months. During this time, they visit the study site about 12 times. Where possible, about 4 of the 12 visits can be done at the participant's home instead of the study site. The trial staff may also contact the participants by phone or video call.

Participants collect urine samples at home. These samples are then analysed to assess kidney function. At the end of the trial the results are compared between the different groups. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients of legal adult age (according to local legislation) and aged ≥ 18 years at time of consent.
* estimated Glomerular Filtration Rate (eGFR, Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 30 and < 90 mL/min/1.73 m2 at Visit 1 by central laboratory analysis.
* Urine Albumin Creatinine Ratio (UACR) ≥ 200 and < 5,000 mg/g in spot urine (midstream urine sample) by central laboratory analysis at Visit 1.1
* If the patient is taking any of the following medications they should be on a stable dose for at least 4 weeks prior to visit 1 and until first randomisation prior to run-in with no planned change of the therapy during the trial: anti-hypertensives, Nonsteroidal Anti-Inflammatory Drugs (NSAIDs), endothelin receptor antagonists, low dose systemic steroids (e.g. prednisolone ≤10 mg or equivalent).
* Treatment with a clinically appropriate, stable dose of either Angiotensin-Converting Enzyme Inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) (but not both together), for ≥ 4 weeks prior to visit 1 and until first randomisation with no planned change of the therapy during the trial.
* In the Investigator's opinion, any kind of diagnosed chronic kidney disease (Diagnosis can be reached by standard clinical method, no biopsy required). Patients with diabetic kidney disease must have type 2 diabetes mellitus and their treatment (including GLP1 receptor agonist) should be unchanged or changes deemed minor (according to investigator's judgement) within 4 weeks prior to Visit 1 and until first randomisation.
* Glycated Haemoglobin (HbA1c) < 10.0% at Visit 1 measured by the central laboratory.
* Serum potassium ≤ 4.8 mmol/L at Visit 1 measured by the central laboratory.
* Seated Systolic Blood Pressure (SBP) ≥ 110 and ≤ 160 mmHg and Diastolic Blood Pressure (DBP) ≥ 65 and ≤ 110 mmHg at Visit 1 (mean values from three Blood Pressure (BP) measurements) and optimised anti-hypertensive treatment according to local standard of care and investigator's judgement.
* Body Mass Index (BMI) ≥ 18.5 and < 50 kg/m2 at Visit 1.
* Women of child-bearing potential2 (WOCBP) must be ready and able to use highly effective methods of birth control. Such methods should be used throughout the trial. Men must be vasectomised or willing and able to use a condom if their partner is a WOCBP.

Additional inclusion criteria to be assessed before second randomisation (start of Treatment Period):

* Serum potassium ≤ 4.8 mmol/L measured by local or central laboratory within 7 days prior to randomisation to the Treatment Period.
* eGFR (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 20 mL/min/1.73 m2 measured by local or central laboratory within 7 days prior to randomisation to the Treatment Period.

Exclusion criteria

* Treatment with inhibitors of aldosterone mediated effects (e.g., mineralocorticoid receptor antagonists such as spironolactone), or intake of other potassium sparing diuretics (e.g., amiloride) within 7 days prior to first randomisation or planned during trial treatment phase.
* Treatment with other Renin Angiotensin Aldosterone System (RAAS) interventions (apart from either Angiotensin-Converting Enzyme Inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB)) within 4 weeks prior to Visit 1 and throughout screening or planned during the trial. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial are also excluded.
* Type 1 diabetes mellitus, or history of other autoimmune causes of diabetes mellitus (e.g. Latent Autoimmune Diabetes (LADA))
* Patients at increased risk of ketoacidosis in the opinion of the investigator.
* Currently receiving Sodium-glucose cotransporter (SGLT)-2 or SGLT-1/2 inhibitor or planned initiation during the trial.

Further criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (203):
- United States (41):
  - Aventiv Research Inc., Mesa, Arizona
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - Clearview Medical Research, LLC, Canyon Country, California
  - Pacific Renal Associates, Long Beach, California
  - Amicis Research Center, Northridge, California
  - Valley Clinical Trials, Inc., Northridge, California
  - California Kidney Specialists, San Dimas, California
  - Colorado Kidney Care, Denver, Colorado
  - Clinical Research of Brandon LLC, Brandon, Florida
  - Horizon Research Group, Coral Gables, Florida
  - Elixia Fort Lauderdale, LLC, Fort Lauderdale, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Total Research Group, LLC, Miami, Florida
  - Horizon Research Group, LLC, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Elixia Tampa, LLC, Temple Terrace, Florida
  - Boise Kidney and Hypertension PLLC, Nampa, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Aa Mrc Llc, Flint, Michigan
  - Elite Research Center, LLC, Flint, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Forte Family Practice, Las Vegas, Nevada
  - New Mexico Clinical Research and Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Triad Internal Medicine, Asheboro, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Diabetes & Endocrinology Associates of Stark County, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Elixia Upland, LLC, Upland, Pennsylvania
  - Monument Health, Rapid City, South Dakota
  - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - Academy Of Diabetes, Thyroid And Endocrine, PA, El Paso, Texas
  - PrimeCare Medical Group, Houston, Texas
  - P&I Clinical Research, LLC, Lufkin, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Providence Medical Research Center, Spokane, Washington
  - Universal Research Group, LLC, Tacoma, Washington
- Argentina (8):
  - CIMEL centro de Investigaciones Médicas Lanús, Buenos Aires
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Glenny Corp. S.A. Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Instituto Privado de Investigaciones Clínica Córdoba S.A., Córdoba
  - Centro de Salud Renal Junín, Junín
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto Médico Catamarca - IMEC, Rosario
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (3):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Monash University, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Belgium (5):
  - Brussels - UNIV UZ Brussel, Brussels
  - Brussels - UNIV Saint-Luc, Brussels
  - La Louvière - UNIV CHU Tivoli, La Louvière
  - UZ Leuven, Leuven/Vlaams-Brabant
  - Charleroi - UNIV CHU de Charleroi, Lodelinsart
- Brazil (9):
  - Hospital Universitário João de Barros Barreto, Belém
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Fundação Pró Renal Brasil, Curitiba
  - Universidade Federal do Rio Grande do Sul, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - BR Trials, São Paulo
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - Hospital do RIM - UNIFESP, São Paulo
- Bulgaria (4):
  - Medical Center Rusemed, Rousse
  - Robert Koch Clinic Sofia, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
  - MHAT Prof Stoyan Kirkovich AD, Stara Zagora
- Canada (6):
  - The Bailey Clinic, Red Deer, Alberta
  - LMC Clinical Research Inc. (Brampton), Brampton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
  - Shivinder Jolly, Nephrologist, Waterloo, Ontario
  - Recherche GCP Research, Montreal, Quebec
- China (6):
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - The First People's Hospital of Nanning, Nanning
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
- Czechia (4):
  - DIKa centrum s.r.o., Havířov
  - Synexus Czech s.r.o., Prague
  - MILAN KVAPIL s.r.o., Příbram
  - Hospital Slany, Internal Department, Slaný
- Finland (3):
  - Satucon Oy, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital / TYKS, Turku
- Germany (9):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Institut für klinische Forschung und Entwicklung (IKFE) Berlin GmbH, Berlin
  - Cardiologicum Dresden und Pirna, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - DaVita Clinical Research Germany GmbH, Düsseldorf
  - Synexus Clinical Research GmbH, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Synexus Clinical Research GmbH, Leipzig
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Greece (4):
  - General Hospital of Athens "Laiko", Athens
  - "Attiko" Hospital of Athens, Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - Iatriko of Athens Group/ Iatriko of P. Faliro, P. Faliro
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (7):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - DRC Drug Research Ltd, Balatonfüred
  - Synexus Hungary Healthcare Service Ltd., Budapest
  - Semmelweis University, Budapest
  - University Debrecen Hospital, Debrecen
  - Markhot Ferenc Hospital, Eger, Eger
  - BKS Research Ltd, Hatvan
- India (10):
  - Government Medical College & Hospital, Aurangabad
  - SMS Medical College and HospitaL, Jaipur
  - Jaipur National University Institute for Medical Science & Research Centre, Jaipur
  - Ganesh Shankar Vidyarthi Memorial Medical College, Kanpur
  - K R Hospital Mysore Medical College and Research Centre, Mysore
  - Kingsway Hospitals, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Galaxy Lifecare Services Pvt. Ltd., Varanasi
  - Christian Medical College, Vellore
- Italy (2):
  - A.O. Policlinico Giovanni XXIII di Bari, Bari
  - ASST Papa Giovanni XXIII - A.O. Papa Giovanni XXIII, Bergamo
- Japan (14):
  - Daiyukai Clinic, Aichi, Ichinomiya
  - Meitetsu Hospital, Aichi, Nagoya
  - Nagoya Kyoritsu Hospital, Aichi, Nagoya
  - TOSAKI Clinic for Diabetes and Endocrinology, Aichi, Nagoya
  - National Hospital Organization Takasaki General Medical Center, Gumma, Takasaki
  - Kyoto Okamoto Memorial Hospital, Kyoto, Kuse-gun
  - Ina Central Hospital, Nagano, Ina
  - Suwa Red Cross Hospital, Nagano, Suwa
  - Asano Clinic, Saitama, Kawagoe
  - Omihachiman Community Medical Center, Shiga, Omihachiman
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
  - Miho Clinic, Tokyo, Shinagawa-ku
  - Yamaura Medical Clinic, Ueda, Nagano
- Malaysia (6):
  - Hospital Selayang, Batu Caves
  - University Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Klinik Kesihatan Mahmoodiah, Johor Bahru
  - Tuanku Fauziah Hospital, Kangar
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kota Bharu
  - Hospital Seri Manjung, Seri Manjung
- Mexico (7):
  - Centro de Investigacion Cardiometabolica de Aguascalientes, Aguascalientes
  - Unidad de Investigación Clinica y Atencion Medica HEPA SC, Guadalajara
  - Centro Mexicano de Desarrollo de Estudios Clínicos SA -CEMDEC, México
  - Clinstile S.A. de C.V., México
  - CEDOPEC-Ctro Esp en Diab, Obesidad y Prev de Enf Cardiovasc, México
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
- Norway (2):
  - Akershus Universitetssykehus HF, Nordbyhagen
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
- Philippines (7):
  - Norzel Medical and Diagnostic Clinic, Cebu City
  - Davao Doctors Hospital, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - Institute for Studies on Diabetes Foundation Inc., Marikina City
  - The Medical City, Pasig
  - Philippine Heart Center, Quezon City
  - Senor Santo Nino Hospital, Tarlac City
- Poland (14):
  - INTERCORE Medical Center, Bydgoszcz
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Katowice
  - Pro Familia Altera, Katowice
  - Synexus Lodz Medical Center, Lodz
  - Clinical Best Solutions, Lublin
  - NZOZ Specialized Ambulance "MEDICA", Lublin
  - Hospitals of Tczew S.A., Pomorskie
  - Omedica Medical Centre, Poznan, Poznan
  - Synexus Poland, Branch in Poznan, Poznan
  - Medical Center HCP Sp. z o.o, Poznan
  - Centrum Medyczne Synexus, Warsaw
  - Barwijuk Clinics, Warsaw
  - Synexus Poland, Branch in Wroclaw, Wroclaw
- Portugal (6):
  - ULS de Almada -Seixal, E. P. E. - Hospital Garcia de Orta, Almada
  - ULS da Região de Aveiro, Aveiro
  - CHLO, EPE - Hospital de Santa Cruz, Carnaxide
  - ULS da Região de Leiria, E.P.E., Leiria
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - ULS de Gaia/Espinho, EPE, Vila Nova de Gaia
- South Africa (8):
  - Iatros International, Bloemfontein
  - Synexus Helderberg Clinical Research Centre, Cape Town
  - TREAD Research, Cape Town
  - Langeberg Clinical Trials, Cape Town
  - Paarl Research Centre, Cape Town
  - Latiff, GHVM, Durban
  - DJW Navorsing, Krugersdorp
  - Synexus Watermeyer Clinical Research Centre, Pretoria
- South Korea (6):
  - Korea University Ansan Hospital, Ansan
  - Chungbuk National University Hospital, Cheongiu
  - Inje University Ilsan Paik Hospital, Goyang
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Público Da Mariña, Burela de Cabo
  - Hospital Universitario Reina Sofía, Córdoba
  - Fundación Jiménez Díaz, Madrid
  - Hospital Puerta de Hierro, Majadahonda
- Sweden (3):
  - Centralsjukhuset, Kristianstad, Kristianstad
  - Universitetssjukhuset, Linköping, Linköping
  - Citydiabetes, Stockholm, Stockholm
- University Hospital of Lausanne, Lausanne, Switzerland
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Once the time frame criteria given under number 4 are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Gashaw IA, Tuttle KR, Monroy Kuhn M, Pleiner S, Delic D, Cronin L, Shah SV, Rossing P. Pharmacodynamics of vicadrostat for aldosterone synthase inhibition in patients with CKD. Eur J Endocrinol. 2026 Jan 6;194(1):46-57. doi: 10.1093/ejendo/lvaf265. PMID 41436034
- [Derived] Tuttle KR, Hauske SJ, Canziani ME, Caramori ML, Cherney D, Cronin L, Heerspink HJL, Hugo C, Nangaku M, Rotter RC, Silva A, Shah SV, Sun Z, Urbach D, de Zeeuw D, Rossing P; ASi in CKD group. Efficacy and safety of aldosterone synthase inhibition with and without empagliflozin for chronic kidney disease: a randomised, controlled, phase 2 trial. Lancet. 2024 Jan 27;403(10424):379-390. doi: 10.1016/S0140-6736(23)02408-X. Epub 2023 Dec 15. PMID 38109916
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial included two randomisations, R1 and R2. At first randomisation R1, patients were 1:1 randomised to a run-in period of 8 weeks and received 10 mg empagliflozin or placebo matching empagliflozin. The run-in period was followed by randomisation R2 at which patients were 1:1:1:1 randomized to a treatment period of 14 weeks to receive one of three doses of BI 690517 or placebo matching BI 690517 in combination with the background medication assigned in the randomized run-in period.
Pre-assignment Details: 2 patients of the arm "Run-in period: Placebo to empagliflozin 10 mg" who did not complete the Run-in period (RP) were mistakenly randomized to the treatment period (TP) but were not treated during the TP with BI 690517 or placebo to BI 690517.
Groups:
- Run-in Period: 10 mg Empagliflozin: Patients received during the run-in period 10 milligrams (mg) of empagliflozin once daily orally for 8 weeks.
- Run-in Period: Placebo to Empagliflozin 10 mg: Patients received during the run-in period placebo matching empagliflozin 10 milligrams (mg) once daily orally for 8 weeks.
- Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517: This arm includes patients who received 10 mg of empagliflozin during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 3 milligrams (mg) of BI 690517 once daily (QD) orally in combination with 10 mg of empagliflozin QD orally. Patients received 3 mg BI 690517 and 10 mg empagliflozin for 14 weeks.
- Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517: This arm includes patients who received 10 mg of empagliflozin during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 10 milligrams (mg) of BI 690517 once daily (QD) orally in combination with 10 mg of empagliflozin QD orally. Patients received 10 mg BI 690517 and 10 mg empagliflozin for 14 weeks.
- Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517: This arm includes patients who received 10 mg of empagliflozin during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 20 milligrams (mg) of BI 690517 once daily (QD) orally in combination with 10 mg of empagliflozin QD orally. Patients received 20 mg BI 690517 and 10 mg empagliflozin for 14 weeks.
- Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517: This arm includes patients who received 10 mg of empagliflozin during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received placebo matching BI 690517 once daily (QD) orally in combination with 10 mg of empagliflozin QD orally. Patients received placebo matching BI 690517 and 10 mg empagliflozin for 14 weeks.
- Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517: This arm includes patients who received placebo matching empagliflozin 10 milligrams (mg) during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 3 mg of BI 690517 once daily (QD) orally in combination with placebo matching empagliflozin 10 mg QD orally. Patients received 3 mg BI 690517 and placebo matching empagliflozin 10 mg for 14 weeks.
- Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517: This arm includes patients who received placebo matching empagliflozin 10 milligrams (mg) during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 10 mg of BI 690517 once daily (QD) orally in combination with placebo matching empagliflozin 10 mg QD orally. Patients received 10 mg BI 690517 and placebo matching empagliflozin 10 mg for 14 weeks.
- Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517: This arm includes patients who received placebo matching empagliflozin 10 milligrams (mg) during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received 20 mg of BI 690517 once daily (QD) orally in combination with placebo matching empagliflozin 10 mg QD orally. Patients received 20 mg BI 690517 and placebo matching empagliflozin 10 mg for 14 weeks.
- Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517: This arm includes patients who received placebo matching empagliflozin 10 milligrams (mg) during the run-in period and met the eligibility criteria to enter the treatment period.
  In the treatment period patients received placebo matching BI 690517 once daily (QD) orally in combination with placebo matching empagliflozin 10 mg QD orally. Patients received placebo matching BI 690517 and placebo matching empagliflozin 10 mg for 14 weeks.
Period: Run-in Period
Arm/Group | Run-in Period: 10 mg Empagliflozin | Run-in Period: Placebo to Empagliflozin 10 mg | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Started (Randomised to Run-in period) | 356 | 358 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated With Empagliflozin 10 mg or Placebo Matching Empagliflozin 10 mg | 356 | 357 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 332 | 330 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 24 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other reason but not sponsor termination | 14 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No reason available | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Burden of study procedures | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Change of residence | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Completed RP and Randomized to TP
Arm/Group | Run-in Period: 10 mg Empagliflozin | Run-in Period: Placebo to Empagliflozin 10 mg | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Started (Completed planned Run-in period) | 332 | 330 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Randomised to Treatment period) | 298 | 286 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 34 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet additional inclusion/exclusion criteria for Treatment Period | 34 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Patients Starting the Treatment Period
Arm/Group | Run-in Period: 10 mg Empagliflozin | Run-in Period: Placebo to Empagliflozin 10 mg | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Started | 298 | 288 (2 participants of this arm who did not complete the Run-in period were randomized mistakenly to the Treatment Period. Therefore 2 milestones below were added.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Did Not Complete the run-in Period and Was Randomized to Treatment Period | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed run-in Period and Randomized to Treatment Period | 298 | 286 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 298 | 288 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Run-in Period: 10 mg Empagliflozin | Run-in Period: Placebo to Empagliflozin 10 mg | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Started (Randomised to Treatment period) | 0 (Patients who received empagliflozin in the Run-in Period and met the eligibility criteria to enter the Treatment Period were randomised equally into one of four parallel dose groups in a 1:1:1:1 ratio to receive one of 3 doses of BI 690517 (3 mg QD, 10 mg QD or 20 mg QD) in combination with empagliflozin, or empagliflozin alone (empagliflozin plus placebo matching to BI 690517).) | 0 (Patients who received placebo in the Run-in Period were randomised equally into one of four parallel dose groups in a 1:1:1:1 ratio to receive one of 3 doses of BI 690517 (3 mg QD, 10 mg QD or 20 mg QD) or placebo (placebo to empagliflozin placebo matching to BI 690517).) | 76 | 74 | 74 | 74 | 71 | 72 | 72 | 73
Treated With BI 690517 or Placebo Matching BI 690517 | 0 | 0 | 76 | 73 | 74 | 74 | 70 | 71 | 72 | 73
Completed (Completed planned treatment with BI 690517 or placebo matching BI 690517) | 0 | 0 | 63 | 50 | 55 | 58 | 61 | 54 | 48 | 66
Not Completed | 0 | 0 | 13 | 24 | 19 | 16 | 10 | 18 | 24 | 7
Not completed — Reason missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other but not sponsor termination | 0 | 0 | 8 | 6 | 6 | 7 | 5 | 8 | 7 | 2
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — No reason available | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Burden of study procedures | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Change of residence | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 16 | 12 | 6 | 4 | 8 | 16 | 5
Not completed — Not treated with study drug | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): This patient set included all entered and randomised patients based on the treatment groups they were randomised to at the randomisation prior to the treatment period (i.e. at second randomisation (R2)), regardless of being treated by BI 690517 or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517 | Total
Number analyzed (Participants) | 76 | 74 | 74 | 74 | 71 | 72 | 72 | 73 | 586
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (11.2) | 64.4 (12.3) | 61.8 (12.2) | 63.4 (10.3) | 64.4 (11.8) | 64.8 (9.9) | 64.3 (10.7) | 62.3 (11.4) | 63.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 20 | 31 | 20 | 23 | 27 | 18 | 196
  Male | 49 | 44 | 54 | 43 | 51 | 49 | 45 | 55 | 390
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 21 | 12 | 20 | 22 | 21 | 18 | 24 | 163
  Not Hispanic or Latino | 51 | 53 | 62 | 54 | 49 | 51 | 54 | 49 | 423
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 2 | 2 | 2 | 3 | 1 | 13
  Asian | 17 | 27 | 20 | 19 | 23 | 15 | 19 | 16 | 156
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 9 | 6 | 7 | 10 | 3 | 9 | 9 | 10 | 63
  White | 49 | 35 | 45 | 42 | 42 | 45 | 40 | 44 | 342
  More than one race | 1 | 4 | 1 | 1 | 1 | 1 | 1 | 1 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine Albumin Creatinine Ratio (UACR) at baseline [Mean (Standard Deviation); unit: milligram/gram] — UACR is a ratio between two measured substances i.e., albumine and creatinine and it is calculated as: (Urine albumin (milligram (mg)/deciliter (dL)))/(urine creatinine gram (g)/deciliter (dL))= UACR in mg/g.
  Albuminuria is present when UACR is greater than 30 mg/g and is a marker for chronic kidney disease (CKD).
  UACR measurements were collected on 2 consecutive days at 3 timepoints from Week -2 to Week 0 (i.e. Week 6-8 of Run-in period) for treatment period baseline. Population: Randomised Set (RS): This patient set included all entered and randomised patients based on the treatment groups they were randomised to at the randomisation prior to the treatment period (i.e. at second randomisation (R2)), regardless of being treated by BI 690517 or not.
  Three patients in the RS had missing baseline values for UACR.
  milligram/gram
    number analyzed (Participants) | 76 | 73 | 74 | 74 | 70 | 71 | 72 | 73 | 583
    (all) | 780.3 (828.8) | 740.8 (915.0) | 695.4 (748.0) | 801.4 (1132.3) | 934.0 (1363.6) | 646.2 (685.2) | 785.0 (885.7) | 684.4 (715.1) | 757.9 (930.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Treatment Period Baseline in Log Transformed Urine Albumin Creatinine Ratio (UACR) Measured in First Morning Void (FMV) Urine After 14 Weeks - All Patients
Description: The adjusted mean change (95% confidence interval) in log transformed FMV UACR from baseline at 14 weeks is presented.
  The adjusted means and 95 % confidence intervals were estimated by restricted maximum likelihood-based mixed models for repeated measures ((REML)-based MMRM) which includes the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated UACR measurements from baseline (Week 6,7 or 8 of the Run-in period) and Week 6, Week 10 and Week 12-14 of Treatment period.
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 (3mg QD, 10 mg QD or 20 mg QD) or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (milligram/gram)
Groups:
- 3 mg BI 690517: This arm includes patients who received during the Treatment Period 3 milligram (mg) of BI 690517 + 10 mg Empagliflozin (i.e. arm "Treatment period: 10 mg empagliflozin + 3 mg BI 690517" in the Participant Flow) and patients who received during the Treatment period 3 mg BI 690517 + Placebo matching Empagliflozin 10 mg (i.e. arm "Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517" in the Participant Flow).
- 10 mg BI 690517: This arm includes patients who received during the Treatment Period 10 milligram (mg) of BI 690517 + 10 mg Empagliflozin (i.e. arm "Treatment period: 10 mg empagliflozin + 10 mg BI 690517" in the Participant Flow) and patients who received during the Treatment period 10 mg BI 690517 + Placebo matching Empagliflozin 10 mg (i.e. arm "Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517" in the Participant Flow).
- 20 mg BI 690517: This arm includes patients who received during the Treatment Period 20 milligram (mg) of BI 690517 + 10 mg Empagliflozin (i.e. arm "Treatment period: 10 mg empagliflozin + 20 mg BI 690517" in the Participant Flow) and patients who received during the Treatment period 20 mg BI 690517 + Placebo matching Empagliflozin 10 mg (i.e. arm "Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 690517" in the Participant Flow).
- Placebo to BI 690517: This arm includes patients who received during the Treatment Period Placebo to BI 690517 + 10 mg Empagliflozin (i.e. arm "Treatment period: 10 mg empagliflozin + Placebo to BI 690517" in the Participant Flow) and patients who received during the Treatment period Placebo to BI 690517 + Placebo matching Empagliflozin 10 mg (i.e. arm "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517" in the Participant Flow).
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
log (milligram/gram) | -0.235 [-0.355 to -0.114] | -0.553 [-0.681 to -0.425] | -0.487 [-0.616 to -0.357] | -0.066 [-0.184 to 0.051]
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; The difference of adjusted means and 95 % confidence interval were estimated by restricted maximum likelihood-based mixed models for repeated measures ((REML)-based MMRM) which included the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient; Test type: Other; p = 0.0499, MMRM; Mean Difference (Net) = -0.168, 95% CI 2-sided [-0.337 to -0.000] — Least Squares Mean of "3 mg BI 690517" - Least Squares Mean of "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, MMRM; Mean Difference (Net) = -0.486, 95% CI 2-sided [-0.660 to -0.313] — Least Squares Mean of "10 mg BI 690517" - Least Squares Mean of "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, MMRM; Mean Difference (Net) = -0.421, 95% CI 2-sided [-0.596 to -0.246] — Least Squares Mean of "20 mg BI 690517" - Least Squares Mean of "Placebo to BI 690517"
Statistical Analysis 4: Comparison: 3 mg BI 690517 vs 10 mg BI 690517 vs 20 mg BI 690517 vs Placebo to BI 690517; A flat vs. non-flat dose-response relationship across the 3 doses of BI 690517 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod). MMRM estimates were used as input for the MCP-Mod. MMRM included the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient; Test type: Other — Null hypothesis: The dose-response curve is flat across the 3 BI 690517 doses and the placebo; p = 0.0000, MCPMod Emax model fit — P-value was rounded to four decimal places; Emax model fit assumption: 80% of the maximum effect is achieved at 10 mg
Statistical Analysis 5: Comparison: 3 mg BI 690517 vs 10 mg BI 690517 vs 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 1, analysis 4]; Test type: Other — Null hypothesis: The dose-response curve is flat across the 3 BI 690517 doses and the placebo; p = 0.0000, MCPMod linear model fit — P-value was rounded to four decimal places; Linear model fit assumption: No assumption is needed
Statistical Analysis 6: Comparison: 3 mg BI 690517 vs 10 mg BI 690517 vs 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 1, analysis 4]; Test type: Other — Null hypothesis: The dose-response curve is flat across the 3 BI 690517 doses and the placebo; p = 0.0003, MCPMod exponential model fit; Exponential model fit assumption: 15% of the maximum effect is achieved at 10 mg

2. Primary Outcome: Percent Change of FMV UACR From Baseline to Week 14 Based on Adjusted Median (95% CI) Back Transformed From MMRM Estimate - All Patients
Description: Percent change of first morning void (FMV) urine albumine creatinine ratio (UACR) from baseline to Week 14 based on adjusted median (95% confidence interval (CI)) back transformed from mixed models for repeated measures (MMRM) estimate for all patients is presented.
  Percent change of FMV UACR= (FMV UACR at Week 14-FMV UACR at baseline)*100/(FMV UACR at baseline).
  MMRM included the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent change of FMV UACR
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
percent change of FMV UACR | -20.9 [-29.9 to -10.8] | -42.5 [-49.4 to -34.6] | -38.5 [-46.0 to -30.0] | -6.4 [-16.8 to 5.3]
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; Test type: Other; Median Difference (Net) = -15.5, 95% CI 2-sided [-28.6 to -0.0] — Median of "3 mg BI 690517" - Median of "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; Test type: Other; Median Difference (Net) = -38.5, 95% CI 2-sided [-48.3 to -26.8] — Median of "10 mg BI 690517" - Median of "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; Test type: Other; Median Difference (Net) = -34.3, 95% CI 2-sided [-44.9 to -21.8] — Median of "20 mg BI 690517" - Median of "Placebo to BI 690517"

3. Primary Outcome: Change From Baseline to Week 14 in the Log Transformed FMV UACR - Patients With Background Therapy of Placebo Matching Empagliflozin
Description: The adjusted mean change (95% confidence interval) in log transformed first morning void (FMV) urine albumine creatinine ratio (UACR) from baseline at 14 weeks for patients with background therapy of placebo matching empagliflozin in the Run-in period is presented.
  The adjusted means and 95 % confidence intervals were estimated by restricted maximum likelihood-based mixed models for repeated measures ((REML)-based MMRM) which includes the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: as for outcome 1
Population: All randomised patients to one of 3 doses of BI 690517 (3mg QD, 10 mg QD or 20 mg QD) or placebo matching BI 690517 who received placebo to empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (milligram/gram)
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
log (milligram/gram) | -0.254 [-0.441 to -0.068] | -0.496 [-0.693 to -0.299] | -0.455 [-0.666 to -0.245] | -0.027 [-0.208 to 0.155]
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0867, MMRM; Mean Difference (Net) = -0.227, 95% CI 2-sided [-0.488 to 0.033] — Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517" - Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0007, MMRM; Mean Difference (Net) = -0.469, 95% CI 2-sided [-0.737 to -0.201] — Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517" - Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0027, MMRM; Mean Difference (Net) = -0.429, 95% CI 2-sided [-0.707 to -0.151] — Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 6905177" - Least Squares Mean of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"

4. Primary Outcome: Percent Change of FMV UACR From Baseline to Week 14 Based on Adjusted Median (95% CI) Back Transformed From MMRM Estimate - Patients With Background Therapy of Placebo Matching Empagliflozin
Description: Percent change of first morning void (FMV) urine albumine creatinine ratio (UACR) from baseline to Week 14 based on adjusted median (95% confidence interval (CI)) back transformed from mixed models for repeated measures (MMRM) estimate for patients with background therapy of placebo matching empagliflozin in the Run-in period is presented.
  Percent change of FMV UACR= (FMV UACR at Week 14-FMV UACR at baseline)*100/(FMV UACR at baseline).
  MMRM included the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: percent change of FMV UACR
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
percent change of FMV UACR | -22.4 [-35.6 to -6.5] | -39.1 [-50.0 to -25.8] | -36.6 [-48.6 to -21.7] | -2.6 [-18.8 to 16.8]
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -20.3, 95% CI 2-sided [-38.6 to 3.4] — Median of "Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517" - median of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -37.4, 95% CI 2-sided [-52.2 to -18.2] — Median of "Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517" - median of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -34.9, 95% CI 2-sided [-50.7 to -14.0] — Median of "Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 6905177" - median of "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"

5. Primary Outcome: Change From Baseline to Week 14 in the Log Transformed FMV UACR - Patients With Background Therapy of Empagliflozin
Description: The adjusted mean change (95% confidence interval) in log transformed first morning void (FMV) urine albumine creatinine ratio (UACR) from baseline at 14 weeks for patients with background therapy of empagliflozin in the Run-in period is presented.
  The adjusted means and 95 % confidence intervals were estimated by restricted maximum likelihood-based mixed models for repeated measures ((REML)-based MMRM) which includes the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: as for outcome 1
Population: All randomised patients to one of 3 doses of BI 690517 (3mg QD, 10 mg QD or 20 mg QD) or placebo matching BI 690517 who received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (milligram/gram)
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
log (milligram/gram) | -0.210 [-0.366 to -0.055] | -0.614 [-0.783 to -0.445] | -0.516 [-0.675 to -0.357] | -0.112 [-0.264 to 0.040]
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3737, MMRM; Mean Difference (Net) = -0.098, 95% CI 2-sided [-0.316 to 0.119] — Least Squares Mean of "Treatment period: 10 mg empagliflozin + 3 mg BI 690517" - Least Squares Mean of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, MMRM; Mean Difference (Net) = -0.502, 95% CI 2-sided [-0.730 to -0.275] — Least Squares Mean of "Treatment period: 10 mg empagliflozin + 10 mg BI 690517" - Least Squares Mean of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0004, MMRM; Mean Difference (Net) = -0.404, 95% CI 2-sided [-0.625 to -0.184] — Least Squares Mean of "Treatment period: 10 mg empagliflozin + 20 mg BI 690517" - Least Squares Mean of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"

6. Primary Outcome: Percent Change of FMV UACR From Baseline to Week 14 Based on Adjusted Median (95% CI) of MMRM Estimate - Patients With Background Therapy of Empagliflozin
Description: Percent change of first morning void (FMV) urine albumine creatinine ratio (UACR) from baseline to Week 14 based on adjusted median (95% confidence interval (CI)) back transformed from mixed models for repeated measures (MMRM) estimate for patients with background therapy of empagliflozin in the Run-in period is presented.
  Percent change of FMV UACR= (FMV UACR at Week 14-FMV UACR at baseline)*100/(FMV UACR at baseline).
  MMRM included the fixed effects of treatment at each visit, baseline (continuous) at each visit, and baseline, visit, treatment, background medication (empagliflozin or placebo matching empagliflozin) and randomisation stratum as main effects, as well as random effects of patient.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: percent change of FMV UACR
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
percent change of FMV UACR | -19.0 [-30.6 to -5.4] | -45.9 [-54.3 to -35.9] | -40.3 [-49.1 to -30.0] | -10.6 [-23.2 to 4.1]
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -9.4, 95% CI 2-sided [-27.1 to 12.7] — Median of "Treatment period: 10 mg empagliflozin + 3 mg BI 690517" - median of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -39.5, 95% CI 2-sided [-51.8 to -24.0] — Median of "Treatment period: 10 mg empagliflozin + 10 mg BI 690517" - median of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; Test type: Other; Median Difference (Net) = -33.2, 95% CI 2-sided [-46.5 to -16.8] — Median of "Treatment period: 10 mg empagliflozin + 20 mg BI 690517" - median of "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"

7. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Multiple Imputation
Description: Number of patients with UACR response I is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: UACR measurements from baseline (Week 6,7 or 8 of the Run-in period) and Week 6, Week 10 and Week 12-14 of Treatment period were used for the multiple imputation approach.
Population: Full Analysis Set (FAS): This patient set included all randomised patients who had at least one baseline measurement of UACR at Week -2, -1, or 0 and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 40 | 73 | 66 | 24
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; The odds ratio, 95% confidence interval, and p-value were calculated based on logistic regression of binary outcome adjusting for treatment, and stratification factors as covariates. Randomisation stratification was used, which is based on estimated glomerular filtration rate (eGFR) and urine albumin creatinine ratio (UACR) levels at screening; Test type: Other; p = 0.0136, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.16 to 3.72] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 7.02, 95% CI 2-sided [3.94 to 12.49] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.48, 95% CI 2-sided [3.09 to 9.71] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

8. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Missing as Non-Responder
Description: Number of patients with UACR response I is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 (3mg QD, 10 mg QD or 20 mg QD) or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 40 | 62 | 57 | 23
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0111, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.19 to 3.88] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.33, 95% CI 2-sided [3.49 to 11.49] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.21, 95% CI 2-sided [2.88 to 9.44] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

9. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Week - All Patients - Last Observation on Treatment Carried Forward (LOCF)
Description: Number of patients with UACR response I is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: UACR measurements from baseline (Week 6,7 or 8 of the Run-in period) and Week 6, Week 10 and Week 12-14 of Treatment period were used for the last observation carried forward approach.
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 (3mg QD, 10 mg QD or 20 mg QD) or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Measure: Count of Participants; unit: Participants
Groups:
- BI 690517 3 mg: This arm includes patients who received during the Treatment Period 3 milligram (mg) of BI 690517 + 10 mg Empagliflozin (i.e. arm "Treatment period: 10 mg empagliflozin + 3 mg BI 690517" in the Participant Flow) and patients who received during the Treatment period 3 mg BI 690517 + Placebo matching Empagliflozin 10 mg (i.e. arm "Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517" in the Participant flow).
Arm/Group | BI 690517 3 mg | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 45 | 67 | 73 | 31
Statistical Analysis 1: Comparison: BI 690517 3 mg vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0348, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.04 to 3.09] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.12, 95% CI 2-sided [2.40 to 7.08] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.02, 95% CI 2-sided [2.91 to 8.67] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

10. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Complete Case Analysis
Description: Number of patients with UACR response I is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (i.e. Week 6, 7 or 8 of Run-in period) and one post-baseline measurement at Week 12-14 when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 124 | 107 | 106 | 127
Participants | 40 | 62 | 57 | 23
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0111, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.19 to 3.88] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.33, 95% CI 2-sided [3.49 to 11.49] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.21, 95% CI 2-sided [2.88 to 9.44] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

11. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Placebo Matching Empagliflozin - Multiple Imputation
Description: Number of patients with UACR response I for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: as for outcome 7
Population: All randomised patients to one of 3 doses of BI 690517 or placebo to BI 690517 who received placebo to empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo to BI 690517. The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 19 | 31 | 30 | 10
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0419, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.03 to 5.74] — Odds ratio of "Treatment period: Placebo to empagliflozin 10 mg + 3 mg BI 690517" vs. "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.09, 95% CI 2-sided [2.64 to 14.08] — Odds ratio of "Treatment period: Placebo to empagliflozin 10 mg + 10 mg BI 690517" vs. "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.13, 95% CI 2-sided [2.64 to 14.25] — Odds ratio of "Treatment period: Placebo to empagliflozin 10 mg + 20 mg BI 690517" vs. "Treatment period: Placebo to empagliflozin 10 mg + Placebo to BI 690517"

12. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Placebo Matching Empagliflozin - Missing as Non-Responder
Description: Number of patients with UACR response I for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who received placebo to empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517. The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 19 | 28 | 25 | 9
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0195, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.19 to 7.02] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.38, 95% CI 2-sided [2.65 to 15.35] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0001, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.39, 95% CI 2-sided [2.60 to 15.67] — [estimate comment as in outcome 11, analysis 3]

13. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in FMV Urine of UACR From Treatment Period Baseline to 14 Weeks - Background Therapy of Placebo Matching Empagliflozin - Last Observation on Treatment Carried Forward (LOCF)
Description: Number of patients with UACR response I for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void (FMV) urine of UACR from treatment period baseline to 14 weeks.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: as for outcome 9
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who received placebo to empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517. LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 22 | 31 | 32 | 14
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0767, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.93 to 4.42] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0003, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.11, 95% CI 2-sided [1.89 to 8.91] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0001, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.69, 95% CI 2-sided [2.15 to 10.24] — [estimate comment as in outcome 11, analysis 3]

14. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Placebo Matching Empagliflozin - Complete Case Analysis
Description: Number of patients with UACR response I for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had received placebo matching empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (i.e. Week 6, 7 or 8 of Run-in period) and one post-baseline measurement at Week 12-14 when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 61 | 56 | 50 | 66
Participants | 19 | 28 | 25 | 9
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0195, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.19 to 7.02] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.38, 95% CI 2-sided [2.65 to 15.35] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0001, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.39, 95% CI 2-sided [2.60 to 15.67] — [estimate comment as in outcome 11, analysis 3]

15. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Multiple Imputation
Description: Number of patients with UACR response I for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: as for outcome 7
Population: All randomised patients to of 3 doses of BI 690517 or placebo matching BI 690517 who received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517. The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 21 | 42 | 36 | 14
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.1398, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.82 to 4.04] — Odds ratio of "Treatment period: 10 mg empagliflozin + 3 mg BI 690517" vs. "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 8.42, 95% CI 2-sided [3.73 to 19.02] — Odds ratio of "Treatment period: 10 mg empagliflozin + 10 mg BI 690517" vs. "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other — P-value was rounded to four decimal places; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.98, 95% CI 2-sided [2.28 to 10.90] — Odds ratio of "Treatment period: 10 mg empagliflozin + 20 mg BI 690517" vs. "Treatment period: 10 mg empagliflozin + Placebo to BI 690517"

16. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Missing as Non-Responder
Description: Number of patients with UACR response I for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517. The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 21 | 34 | 32 | 14
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.1884, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.77 to 3.79] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.80, 95% CI 2-sided [2.94 to 15.72] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0003, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.46, 95% CI 2-sided [2.00 to 9.94] — [estimate comment as in outcome 15, analysis 3]

17. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Last Observation on Treatment Carried Forward
Description: Number of patients with UACR response I for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Last observation on treatment carried forward (LOCF) uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: as for outcome 9
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 23 | 36 | 41 | 17
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.2140, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.76 to 3.46] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0003, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.13, 95% CI 2-sided [1.93 to 8.85] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.43, 95% CI 2-sided [2.52 to 11.71] — [estimate comment as in outcome 15, analysis 3]

18. Secondary Outcome: UACR Response I, Defined as Decrease of at Least 30% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Complete Case Analysis
Description: Number of patients with UACR response I for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response I was defined as decrease of at least 30% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (i.e. Week 6, 7 or 8 of Run-in period) and one post-baseline measurement at Week 12-14 when patients were still on treatment with BI 690517 or placebo matching BI 690517.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 51 | 56 | 61
Participants | 21 | 34 | 32 | 14
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.1884, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.77 to 3.79] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.80, 95% CI 2-sided [2.94 to 15.72] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0003, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.46, 95% CI 2-sided [2.00 to 9.94] — [estimate comment as in outcome 15, analysis 3]

19. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients -Multiple Imputation
Description: Number of patients with UACR response II is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 week. The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: as for outcome 7
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 68 | 82 | 81 | 46
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0024, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.32 to 3.61] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.05, 95% CI 2-sided [2.39 to 6.86] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.87, 95% CI 2-sided [2.29 to 6.55] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

20. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Missing as Non-Responder
Description: Number of patients with UACR response II is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 67 | 71 | 70 | 44
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0019, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.35 to 3.77] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.81, 95% CI 2-sided [2.20 to 6.59] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.67, 95% CI 2-sided [2.12 to 6.35] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

21. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Last Observation on Treatment Carried Forward (LOCF)
Description: Number of patients with UACR response II is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: as for outcome 9
Population: Full Analysis Set (FAS): This patient set included all randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6, 7 or 8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 128 | 121 | 121 | 133
Participants | 67 | 87 | 85 | 53
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0418, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.02 to 2.74] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.91, 95% CI 2-sided [2.30 to 6.65] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.58, 95% CI 2-sided [2.11 to 6.05] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

22. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - All Patients - Complete Case Analysis
Description: Number of patients with UACR response II is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg BI 690517 | 10 mg BI 690517 | 20 mg BI 690517 | Placebo to BI 690517
Number analyzed (Participants) | 124 | 107 | 106 | 127
Participants | 67 | 71 | 70 | 44
Statistical Analysis 1: Comparison: 3 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0019, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.35 to 3.77] — Odds ratio of "3 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 2: Comparison: 10 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.81, 95% CI 2-sided [2.20 to 6.59] — Odds ratio of "10 mg BI 690517" vs. "Placebo to BI 690517"
Statistical Analysis 3: Comparison: 20 mg BI 690517 vs Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.67, 95% CI 2-sided [2.12 to 6.35] — Odds ratio of "20 mg BI 690517" vs. "Placebo to BI 690517"

23. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Placebo Matching Empagliflozin - Multiple Imputation
Description: Number of patients with UACR response II for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: as for outcome 7
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 33 | 35 | 39 | 22
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0285, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.09 to 4.45] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0038, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.41 to 5.96] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0002, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.97 to 8.72] — [estimate comment as in outcome 11, analysis 3]

24. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Placebo Matching Empagliflozin - Missing as Non-Responder
Description: Number of patients with UACR response II for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 32 | 32 | 32 | 20
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0116, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.23 to 5.31] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0032, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.46 to 6.52] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0004, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.07, 95% CI 2-sided [1.86 to 8.91] — [estimate comment as in outcome 11, analysis 3]

25. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in FMV Urine of UACR From Treatment Period Baseline to 14 Weeks - Background Therapy of Placebo Matching Empagliflozin - Last Observation on Treatment Carried Forward (LOCF)
Description: Number of patients with UACR response II for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void (FMV) urine of UACR from treatment period baseline to 14 weeks.
  LOCF uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 65 | 61 | 59 | 69
Participants | 28 | 41 | 41 | 25
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.4092, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.67 to 2.69] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0005, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.77 to 7.58] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0002, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.04, 95% CI 2-sided [1.92 to 8.49] — [estimate comment as in outcome 11, analysis 3]

26. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Multiple Imputation
Description: Number of patients with UACR response II for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Time Frame: as for outcome 7
Population: All randomised patients to one of 3 doses of BI 690517 or placebo matching BI 690517 who received empagliflozin during the Run-in Period and who had at least one baseline measurement of UACR at Week -2, -1, or 0 (Week 6,7,8 of the Run-in Period) and at least one post-baseline measurement when patients were still on treatment with BI 690517 or placebo matching BI 690517. The multiple imputation filled in missing values at Week 14 based on other data observed in the same patient using regression.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 35 | 47 | 42 | 24
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0348, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.06 to 4.43] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0000, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 6.08, 95% CI 2-sided [2.73 to 13.57] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0007, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.58, 95% CI 2-sided [1.71 to 7.52] — [estimate comment as in outcome 15, analysis 3]

27. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Missing as Non-Responder
Description: Number of patients with UACR response II for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  The missing as non-responder imputes patients with missing Week 14 data as non-responders.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 35 | 39 | 38 | 24
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0578, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.98 to 4.14] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0001, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.12, 95% CI 2-sided [2.23 to 11.78] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0022, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.54 to 7.16] — [estimate comment as in outcome 15, analysis 3]

28. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Last Observation on Treatment Carried Forward
Description: Number of patients with UACR response II for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Last observation on treatment carried forward (LOCF) uses the last value observed on treatment to substitute all missing values until Week 14.
Time Frame: as for outcome 9
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 60 | 62 | 64
Participants | 39 | 46 | 44 | 28
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0342, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.06 to 4.44] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0003, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.23, 95% CI 2-sided [1.93 to 9.24] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0023, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.52 to 6.73] — [estimate comment as in outcome 15, analysis 3]

29. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks -Patients With Background Therapy of Placebo Matching Empagliflozin - Complete Case Analysis
Description: Number of patients with UACR response II for patients with background therapy of placebo matching empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
Number analyzed (Participants) | 61 | 56 | 50 | 66
Participants | 32 | 32 | 32 | 20
Statistical Analysis 1: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0116, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.23 to 5.31] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0032, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.46 to 6.52] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 vs Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0004, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 4.07, 95% CI 2-sided [1.86 to 8.91] — [estimate comment as in outcome 11, analysis 3]

30. Secondary Outcome: UACR Response II, Defined as Decrease of at Least 15% Absolute Change in First Morning Void Urine of UACR From Treatment Period Baseline to 14 Weeks - Patients With Background Therapy of Empagliflozin - Complete Case Analysis
Description: Number of patients with UACR response II for patients with background therapy of empagliflozin in the Run-in period is reported. UACR response II was defined as decrease of at least 15% absolute change in First Morning Void urine of UACR from treatment period baseline to 14 weeks.
  Complete case analysis used patients with both baseline and Week 14 data available.
Time Frame: At baseline (Week 6,7 or 8 of the Run-in period) and at Week 12-14 of the Treatment Period.
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517
Number analyzed (Participants) | 63 | 51 | 56 | 61
Participants | 35 | 39 | 38 | 24
Statistical Analysis 1: Comparison: Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0578, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.98 to 4.14] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0001, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 5.12, 95% CI 2-sided [2.23 to 11.78] — [estimate comment as in outcome 15, analysis 2]
Statistical Analysis 3: Comparison: Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 vs Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0022, Regression, Logistic — P-value was rounded to four decimal places; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.54 to 7.16] — [estimate comment as in outcome 15, analysis 3]

ADVERSE EVENTS:
Time Frame: Run-in period: From first study drug administration in the run-in period until end of the residual effect period (REP) (i.e., 7 days), up to 9 weeks. Treatment period: From first study drug administration in the treatment period until end of REP (i.e. 7 days), up to 15 weeks. All-Cause Mortality for treatment period: From study drug administration in the treatment period until end of the follow-up period, up to 18 weeks. Continues in the description.
Description: Patients with treatment-emergent adverse events starting during overlapping run-in residual effect period and treatment period are counted in both the run-in period and treatment period.
  Run-in treated set: All randomised patients of the Run-in Period who were documented to have taken at least one dose of empagliflozin or placebo.
  Treated set: All patients who received at least one dose of BI 690517 or placebo matching BI 690517.
Arm/Group | Run-in Period: 10 mg Empagliflozin | Run-in Period: Placebo to Empagliflozin 10 mg | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517
All-Cause Mortality (participants affected / at risk) | 0/356 | 2/357 | 1/76 | 1/73 | 0/74 | 2/74 | 0/70 | 1/71 | 1/72 | 0/73
Serious Adverse Events (participants affected / at risk) | 9/356 | 20/357 | 4/76 | 7/73 | 5/74 | 7/74 | 3/70 | 4/71 | 6/72 | 3/73
Other Adverse Events (participants affected / at risk) | 17/356 | 15/357 | 11/76 | 20/73 | 19/74 | 13/74 | 15/70 | 16/71 | 25/72 | 9/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: 10 mg Empagliflozin (N=356) | Run-in Period: Placebo to Empagliflozin 10 mg (N=357) | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 (N=76) | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 (N=73) | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 (N=74) | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 (N=74) | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 (N=70) | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 (N=71) | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 (N=72) | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517 (N=73)
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcapsular renal haematoma (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coeliac artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: 10 mg Empagliflozin (N=356) | Run-in Period: Placebo to Empagliflozin 10 mg (N=357) | Treatment Period: 10 mg Empagliflozin + 3 mg BI 690517 (N=76) | Treatment Period: 10 mg Empagliflozin + 10 mg BI 690517 (N=73) | Treatment Period: 10 mg Empagliflozin + 20 mg BI 690517 (N=74) | Treatment Period: 10 mg Empagliflozin + Placebo to BI 690517 (N=74) | Treatment Period: Placebo to Empagliflozin 10 mg + 3 mg BI 690517 (N=70) | Treatment Period: Placebo to Empagliflozin 10 mg + 10 mg BI 690517 (N=71) | Treatment Period: Placebo to Empagliflozin 10 mg + 20 mg BI 690517 (N=72) | Treatment Period: Placebo to Empagliflozin 10 mg + Placebo to BI 690517 (N=73)
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 1 | 1 | 4 | 4 | 2 | 1 | 3 | 2
Cortisol decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 4 | 2 | 0
Glomerular filtration rate decreased (Investigations) | 4 | 1 | 4 | 8 | 7 | 2 | 1 | 7 | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 8 | 5 | 11 | 7 | 5 | 8 | 7 | 17 | 4
Hypotension (Vascular disorders) | 2 | 0 | 0 | 4 | 2 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05182840/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT05182840/SAP_001.pdf